CLINICAL TRIAL: NCT03969069
Title: Improving the Assessment of Faecal Incontinence: Which Patient Groups Would Benefit From Assessment With Multiple Array Probe Leiden (MAPLe)?
Brief Title: Assessment of Faecal Incontinence With MAPLe
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College London Hospitals (Other)
Responsible Party: Principal Investigator, Rachael Weatherburn, Research Fellow, University College London Hospitals
Other Study IDs: 119731
Record Dates: First submitted 2019-02-13; First posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Faecal Incontinence; Fecal Incontinence; Faecal Incontinence With Faecal Urgency
Keywords: Adult; Human; Cohort
MeSH Terms: conditions — Encopresis; Fecal Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (4):
- Fistula/chronic perianal conditions: Participants symptomatic of FI with chronic perianal disease
  Interventions: Device: MAPLe
- Obstetric injury <12 months: Participants symptomatic of FI < 12 months following obstetric injury.
  Interventions: Device: MAPLe
- Obstetric injury >12 months: Participants symptomatic of FI >12 months following obstetric injury.
  Interventions: Device: MAPLe
- Neurogenic: Participants symptomatic of FI with evidence/history of neurological condition.
  Interventions: Device: MAPLe

INTERVENTIONS:
Device: MAPLe — Additional assessment with MAPLe

SUMMARY:
Faecal incontinence (FI) is the involuntary passage of gas, liquid or solid stool and is experienced by an estimated 1-10% of the population. The symptom is multifactorial and associated with many medical conditions and diseases. The symptom is investigated using structural and functional testing of the pelvic floor. Current investigation techniques have poor correlation between symptom severity and investigation results. These techniques are unable to provide prognostic outcomes, resulting in undirected referrals for treatment based on symptoms alone. This study aims to improve the assessment of FI through additional testing using Multiple Array Probe Leiden (MAPLe). This is a non-invasive medically certified device that detects the electromyography of the pelvic floor, how muscles respond to voluntary nervous stimulus, to identify areas of weakness.

The aim of this study is firstly to identify which patient groups benefit from additional testing with MAPLe, and secondly to identify if directed treatment has been achieved.

The study will take place across two NHS trusts, both with specialist pelvic floor services. Participants referred to each trust with FI who meet the inclusion/exclusion criteria will be recruited from designated pelvic floor clinics and referrals for anorectal physiology (ARP). Each participant will undergo routine anorectal physiological assessment with Anal Ultrasound (AUS) and High Resolution Anal Manometry (HRAM) and additional assessment with MAPLe. Participation is complete unless treatment has been advised, these participants will undergo repeat assessment with MAPLe at 6 months. Average participation will be 12 months.

The results will be analysed to identify non-inferiority of MAPLe vs current techniques using Bland Altman method. Regression and correlation studies will be performed to identify which groups have benefited from assessment with MAPLe. An expert panel of specialists in the field of pelvic floor will be convened to determine the clinical utilisation of MAPLe.

DETAILED DESCRIPTION:
This is cohort study of participants with symptoms of faecal incontinence. The study will take place across two hospital trusts, Ashford and St Peter's NHS Foundation Trust (ASPH) and University Hospital London Hospitals NHS Foundation Trust (UCLH). These trusts have been selected as both provide specialist pelvic floor services and have the facilities required to meet the needs of the study and follow up required by the participants. The use of two sites aims to increase the yield and diversity of participants.

Referrals to each trust are triaged by the overseeing consultant. Potential participants for the study will be identified. At ASPH suitable referrals will be tracked to a dedicated pelvic floor clinic run by a trial representative with medical training. Participants who meet the inclusion/exclusion criteria will be offered a patient information sheet and given an appointment in a dedicated anorectal physiology session (ARP). At UCLH suitable referrals will be contacted via telephone by the PI, should they wish to enrol they will receive a PIS and given an appointment in a dedicated ARP session. Participants will only be assessed and followed up in their recruiting trust.

All participants will complete an incontinence questionnaire and a quality of life questionnaire. Each participant will attend a designated ARP session. At ASPH this will comprise of the current gold standard, Anal Ultrasound (AUS) and High resolution manometry (HRAM) and additional assessment with MAPLe using a standardised protocol. At UCLH participants will undergo AUS in the radiology department, and HRAM and MAPLe in the GI Physiology unit. Through undertaking all three tests participants will act at their own controls. The results will be made available to their overseeing consultant and discussed at their local MDT. Participant participation will conclude following ARP assessment unless treatment is deemed necessary by their local MDT. These participants will be followed up at 6 months with interval MAPLe assessment and incontinence and quality of life questionnaire.

The results will undergo statistical analysis to determine non-inferiority of MAPLe in assessing FI. For analysis participants will be allocated to the following groups: fistula/chronic perianal conditions, obstetric injury <12 months, obstetric injury >12months, neurogenic. Each group will be analysed using symptoms profile and MAPLe results to identify correlation. Comparison of MAPle results pre and post treatment will determine if targeted treatment has been achieved.

An expert panel of pelvic floor specialists will be formed to determine the additional benefit of MAPLe in a clinical context. The panel will consist of 3-6 specialists within the field. To reduce bias, each specialist will be provided with literature on the background of MAPLe and how to analyse the results. The panellists will receive up to date guideline on the management of FI. The panel will be provided with cases and ARP results to answer the following questions:

Question 1: What is the additional benefit of MAPLe?

* Panellists will be provided with clinical history HRAM and AUS results

  ▪ What is the diagnosis and how will you manage this patient?
* MAPLe results provided

  * Has the management changed?
  * How beneficial on scale 1-10 has the addition been? Question 2 : HRAM and AUS vs MAPLe and AUS
* Panellists will be provided with a series of paired histories set one with HRAM and AUS results, set two with MAPLe and AUS results

  * What is the diagnosis and treatment?
  * How confident do you feel in your diagnosis and treatment for set two? Question 3: MAPLe alone
* Panellists will be provided with history and MAPLe results
* What is the diagnosis and treatment?
* Do you feel enough information is provided by the MAPLe to allow for a management plan?

The outcomes of the expert panel will undergo statistical analysis. determine if there is a perceived benefit.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of faecal incontinence
* Capacity to consent

Exclusion criteria:

* Anal surgery in the last 3 months
* Anal cancer
* Acute/painful perianal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All persons symptomatic of faecal incontinence with the capacity to consent and participate who meet the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-05-30 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Which patient groups benefit from assessment with MAPLe? | 12 months
  Identity correlation between symptom profile and MAPLe results
Non-inferiority testing of MAPLe against current ano-rectal physiological tests. | 12 months
  Blank Altman analysis of MAPLE vs HRAM and MAPLe vs AUS

SECONDARY OUTCOMES:
Has directed treatment been achieved? | 18 months
  Identify EMG activity in participants who underwent treatment, compare with pre-treatment EMG

CONTACTS AND LOCATIONS:
Overall Officials: Rachael C Weatherburn, MBChB MRCS, Principal Investigator — Research Fellow
Locations (2):
- United Kingdom (2):
  - St Peter's Hospital, Chertsey, Surrrey
  - University College Hospital, London

IPD SHARING:
Plan to Share IPD: No
Student research project, data will not be shared.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/69/NCT03969069/Prot_SAP_000.pdf